CLINICAL TRIAL: NCT04228094
Title: Development and Assesment of TDApp1 an eHelath Tool to Make Participatory, Patient-centred and Automated Therapeutic Recommendations for Patients With Attention Deficit Hyperactivity Disorder
Brief Title: Assesment of TDApp1 an eHelath Tool to Make Therapeutic Recommendations for Patients With ADHD
Status: Completed | Type: Observational
Sponsor: Universitat de Girona (Other)
Responsible Party: Principal Investigator, Xavier Castells, Development of a web application to formulate participatory, individualized and automated therapeutic recommendations for the treatment of patients with ADHD, Universitat de Girona
Other Study IDs: tdapp1
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Attention Deficit-hyperactivity Disorder
Keywords: eHealth; evidence based medicine; machine learning
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TDApp1: This cohort will use TDApp1: an eHealth tool to formulate participatory, individualized and automated therapeutic recommendations for patients with Attention Deficit Hyperactivity Disorder
  Interventions: Other: TDApp1: an eHealth intervention

INTERVENTIONS:
Other: TDApp1: an eHealth intervention — TDApp1 is a tool that uses GRADE heuristics to formulate participatory, individualized and automated therapeutic recommendations for patients with Attention Deficit Hyperactivity Disorder

SUMMARY:
This is a 3-week open label, one group study to determine the agreement between the pharmacological treatment recommended by TDApp1 and the interventions recommended by relevant clinical practice guidelines.

DETAILED DESCRIPTION:
Clinical practice guidelines (CPGP) allow optimizing medical decisions and health care based on the best evidence available. Nevertheless, CPGs have several limitations. First, many GPC are outdated shortly after their publication. Second, CPG recommendations are often not applicable to many patients treated in clinical practice. Most CPGs do not make recommendations for patients with a mild disorder or for complex patients with comorbiditie. Another limitation is that patients involvement in CPGs development is still poor.

We aim to develop and assess TDApp1: an eHealth tool to formulate participatory, individualized and automated therapeutic recommendations for patients with Attention Deficit Hyperactivity Disorder.

A 3-week, one group, open label study will be conducted. Fifty-five patients aged 6-65 with ADHD will use TDApp1. The therapeutic recommendations made by the TDApp1 and by relevant CPG will be compared. Concordance in the recommendations will be studied. Effectiveness, safety, changes in physical activity and satisfaction will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 6-65
* A diagnosis of DSM-V ADHD based on clinical assessment

Exclusion Criteria:

* Patients under adequate therapeutic treatment or requiring minor adjustments
* Patients lacking an electronic device (mobile phone, tablet,...) with internet access

Ages: 6 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: ADHD patients will be recruited from specialiazed setting.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Treatment recommended/prescribed | 4 days
  Treatment recommended/prescribed consists on the treatment recommended to the patient with ADHD by TDApp1 and the actual treatment prescribed by the investigator to this patient.

SECONDARY OUTCOMES:
Patient/parent satisfaction with the participation in the health decision-making process | 3 weeks
  Satisfaction of the patients or their parents with their participation in the health decision-making process. This outcome will be collected by means of visual analogic scale that has been developed for this study. Score ranges from 1 to 9. Higher scores indicate greater satisfaction.
Patient/parent satisfaction with TDApp1 | 3 weeks
  The satisfaction of the patients or their parents with the educational material provided, and the usability and simplicity of TDApp1. This outcome will be collected by means of visual analogic scale that has been developed for this study. Score ranges from 1 to 9. Higher scores indicate greater satisfaction.
ADHD symptom severity | 3 weeks
  ADHD symptom severity will be assessed with the self-rated, 18-item, DSM V (in children and adolescents) or IV-TR (in adults) -based Rating Scale. Total score ranges from 0 to 54. Higher total scores indicate greater illness severity.
Adverse events | 3 weeks
  The incidence of adverse events will be collected by means of a questionnaire
Patient/parent satisfaction with the treatment prescribed | 3 weeks
  Satisfaction of the patients or their parents with the prescribed treatment. This outcome will be collected by means of visual analogic scale that has been developed for this study. Score ranges from 1 to 9. Higher scores indicate greater satisfaction.
Physical activity | 3 weeks
  The physical activity will be measured by means of ActiGraph wGT3X-BT that records continuous physical activity and sleep/wake information.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Castells, MD, PhD, Principal Investigator — Universitat de Girona
Locations (1):
- Institut d'Assitència Sanitària, Girona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided